CLINICAL TRIAL: NCT06068114
Title: Detailed Assessment of Gastric Functions in Patients With Diabetes Mellitus
Brief Title: Gastric Pathophysiology in Diabetes
Acronym: DiaFLIP
Status: Recruiting | Type: Observational
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Collaborators: Poliklinika Agel, Dopravni zdravotnictvi a.s. (Other)
Responsible Party: Principal Investigator, Doc. (Ass. prof.) Jan Martinek, MD, PhD, AGAF, Prof. Jan Martínek, MD, PhD, AGAF, Institute for Clinical and Experimental Medicine
Other Study IDs: DiaFLIP
Record Dates: First submitted 2023-09-26; First posted 2023-10-05 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Functional Dyspepsia; Gastroparesis; Healthy
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Gastroparesis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetic patients: Either type I or type II diabetes mellitus, possibly also suffering from functional dyspepsia or gastroparesis
- Healthy controls

SUMMARY:
This is a comprehensive pathophysiological study assessing various gastric functions in patients with diabetes mellitus. The investigators aim to examine the stomach with various measurement devices to gain information about its different functions and malfunctions. After the initial measurements, the examinations will be repeated after a year in each patient. Changes in the measurement values will be examined and their relations to each other and to the overall health of the patients will be investigated.

For example it is hypothesised that diabetic patients also suffering from functional dyspepsia or gastroparesis will also show some changes in the function of the pyloric muscle.

ELIGIBILITY:
Inclusion Criteria (diabetic group):

* Diabetes mellitus type I or II, minimal duration of the disease 3 years, minimal duration of specific treatment (drugs, insulin) 2 years

Exclusion Criteria (diabetic group):

* Diabetes mellitus type II being treated with a diet only
* Severe acute decompensation of diabetes (uncontrolled diabetes) necessitating hospitalization
* Concomitant treatment with more than one prokinetic agent
* Active treatment with opioids or a history of treatment with opioids within 12 months before enrolment
* Previous esophageal or major gastric surgery (e.g. esophageal myotomy, esophagectomy, antireflux surgery, Billroth I or II gastric resection, gastric pull-through, pyloromyotomy, pyloroplasty, gastric electrical stimulation)
* Organic pyloric (or intestinal) obstruction (fibrotic stricture, etc.)
* Severe coagulopathy
* Esophageal or gastric varices and /or portal gastropathy
* Advanced liver cirrhosis
* Pregnancy or puerperium
* Malignant or pre-malignant gastric diseases (dysplasia, gastric cancer, GIST): patients with a history of such disease after its cure are eligible for enrolment
* The presence of a rumination syndrome or eating disorders (anorexia nervosa, bulimia). In case of doubts, a psychiatric examination will be performed.
* Systemic connective tissue disorder
* Inability to obtain informed consent
* Any other condition, which in the opinion of the investigator would interfere with study requirements

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Diabetic patients treated in any of the participating centers.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-10-05 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Pyloric distensibility | At baseline and after 12 months
  Pyloric distensibility measured by impedance planimetry (EndoFLIP device)

SECONDARY OUTCOMES:
GCSI score | At baseline and after 6 and 12 months
  Gastroparesis Cardinal Symptom Index questionnaire: The score ranges from 0 to 5 for each symptom (9 questions) and these are averaged into subscores and into a total score (also ranging from 0 to 5). Higher scores indicate more severe symptoms.
PAGI-SYM score | At baseline and after 6 and 12 months
  Patient Assessment of Gastrointestinal Disorders Symptom Severity Index questionnaire: The score ranges from 0 to 5 for each symptom (20 questions) and these are averaged into subscores and into a total score (also ranging from 0 to 5). Higher scores indicate more severe symptoms.
PAGI-QoL score | At baseline and after 6 and 12 months
  Patient Assessment of Upper Gastrointestinal Disorders - Quality of Life questionnaire: The score ranges from 0 to 5 for each symptom (30 questions) and these are averaged into subscores and into a total score (also ranging from 0 to 5). Higher scores indicate lower quality fo life.
Gastric emptying by scintigraphy | At baseline and after 12 months
  Gastric scintigraphy protocol endorsed by both American Neurogastroenterology and Motility Society and American Nuclear Medicine Society will be used to assess gastric emptying with a standard 200 kcal, 2% fat egg-substitute test meal. Gamma camera images will be obtained immediately after meal ingestion and then at 1, 2, 3 and 4 hours. Diagnostic criterion for delayed gastric emptying is defined as the percentage of gastric retention >60% at 2 h or ≥ 10% at 4 h or both. Half-time (T1/2) emptying time will also be calculated. At least 72 hours before gastric emptying test, narcotics and other medications that can interfere with gastric emptying will be discontinued.
Gastric emptying by breath test | At baseline and after 12 months
  Gastric emptying assessed using 13C breath test with octanoic acid. This measurement is an alternative to the measurement of gastric emptying by scintigraphy. The choice depends on the practice in a particular center.
Electrogastrography | At baseline and after 12 months
  Surface electrogastrography (EGG) is a non-invasive method for the evaluation of myoelectric activity of the stomach. Gastric pacemaker generates electrical phenomenon termed "gastric slow waves", which originate in a "pacemaker region" located on the greater curvature near the junction of the fundus and gastric body. EGG recordings will be accomplished by means of EGG Stand (MMS, Enschede, the Netherlands) with a MMS software. Six active self-adhesive electrodes will be placed on the upper part of the abdomen, the 7th electrode (basal) will be placed in the left supraclavicular area. A special abdominal belt (respiratory sensor) will be used to identify possible artefacts due to breathing and body movements . All EGGs will be performed at a lying position in the morning after an overnight fasting. Basal EGG (under fasting condition) will be recorded for 20 minutes. A standard test breakfast will be served afterwards. Postprandial EGG will be recorded for next 40 min.
Autonomic function testing | At baseline and after 12 months
  Autonomic function testing will be performed by the golden standard battery of tests introduced by Ewing. The test involves four phases: (1) resting phase (5 min), (2) deep breathing test (1 min of 0,1 Hz breathing rate), (3) short Valsalva maneuvers (1 min), and (4) standing Tilt test (5 min). An ECG will be recorded during all phases. The Heart rate variability triangular index will be assessed.

CONTACTS AND LOCATIONS:
Locations (5):
- Czechia (4):
  - Nemocnice AGEL Ostrava-Vítkovice a. s., Ostrava
  - University Hospital Ostrava, Ostrava
  - Institute for Clinical and Experimental Medicine, Prague
  - Military University Hospital Prague, Prague
- University Hospital Trnava, Trnava, Slovakia